CLINICAL TRIAL: NCT06858956
Title: Real-World Study of Chidamide Combined With PD-(L)1 Inhibitors and Anti-Angiogenic Therapy for Advanced MSS-Type Colorectal Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, AIPING ZHOU, Doctor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Other Study IDs: CSIIT-Q99
Record Dates: First submitted 2025-02-28; First posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; Bevacizumab; Tyrosine Kinase Inhibitors

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Chidamide, Tucidinostat; PD-1/PD-L1 inhibitor or double antibodies; Bevacizumab or tyrosine kinase inhibitors — Chidamide, Tucidinostat; PD-1/PD-L1 inhibitor or double antibodies; Bevacizumab or tyrosine kinase inhibitors

SUMMARY:
This is an observational , multicenter, real-world study aimed at evaluating the efficacy and safety of the combination of immune checkpoint inhibitors, chidamide and antiangiogenic agents in Microsatellite Stable advanced colorectal cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years, male or female.

Histologically confirmed advanced colorectal cancer with microsatellite stable (MSS)/proficient mismatch repair (pMMR) status confirmed by immunohistochemistry (IHC) or molecular testing.

No restriction on prior immunotherapy or combined anti-angiogenic agents (e.g., bevacizumab or small-molecule TKIs).

ECOG performance status of 0-2.

At least one post-treatment efficacy evaluation.

Life expectancy ≥3 months.

Chidamide treatment duration >3 weeks

Exclusion Criteria:

- 1. Malignancies in other organs or systems, except for cured basal cell/squamous cell skin cancer or cervical carcinoma.

2. Severe comorbidities that may interfere with efficacy or safety analysis. 3. Conditions deemed unsuitable for study inclusion by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Advanced MSS-Type Colorectal Cancer
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
TTF | 24 months

IPD SHARING:
Plan to Share IPD: No